CLINICAL TRIAL: NCT06117228
Title: Gynaecological Follow-up of Women With Down Syndrom Aged 18 to 30 in France
Acronym: Gyn-T21
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_016_Gyn-T21
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Down Syndrome
Keywords: Gynaecological follow-up; down syndrome; women
MeSH Terms: conditions — Down Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women with Down syndrome aged 18 to 30: women aged 18 to 30 with Down syndrome, whether or not they were receiving medical care, who agreed to take part in the study.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Gynaecological check-ups for women are recommended in France. However, some groups of the population are affected by a lack or absence of medical surveillance.

In France, there are one million people with an intellectual disability, including 50,000 with Down syndrome.

Although this disability causes numerous physical and psychological deficits, no gynaecological consequences have yet been demonstrated.

Regular gynaecological check-ups are therefore necessary, according to French recommendations.

However, several studies have shown that women with mental illness receive less or no gynaecological care.

DETAILED DESCRIPTION:
The aim is to describe the gynaecological follow-up of women with Down syndrom in France.

ELIGIBILITY:
Inclusion Criteria:

* women with Down's syndrome,
* aged between 18 and 30,
* whether or not they are being followed up in a medical facility,
* who agree to take part in the study.

Exclusion Criteria:

* women with a disability other than Down's syndrome
* Not agreeing to take part in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with Down syndrome, aged 18 to 30, whether or not they are being followed up in medical facilities in France.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Gynaecological follow-up | Day 0
  Presence or not of gynaecological follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Muller Gaëlle, Principal Investigator — Université de Reims Champagne-Ardenne
Locations (1):
- Ufr Medecine Urca, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided